CLINICAL TRIAL: NCT04837521
Title: Adapting the Unified Protocol to Facilitate Activity in Older Adults
Brief Title: Five Session Unified Protocol for Older Adults With Emotional Distress and Reduced Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108029; 5P30AG064201-03 (NIH); DBSR-11068 (Other Grant/Funding Number: Duke Roybal Center)
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-05

CONDITIONS: Emotional Distress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Phase 1 is Single Group. However, Phase 2 is a parallel comparison of self-guided with therapist-delivered versions of the UP-5
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist Delivered Unified Protocol (Experimental): This is a five session psychotherapy designed to help people with problems such as anxiety and depression.
  Interventions: Behavioral: Unified Protocol
- Self-Guided Unified Protocol (Experimental): This is a five session treatment that patients can complete independently.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — Five session psychotherapy

SUMMARY:
Research suggests older adults report wide-ranging emotional distress (e.g., symptoms of anxiety, depression) that negatively impacts their physical and mental health and is associated with a reduction in daily activity. The overarching goal of this proposal is to adapt an existing evidence-based intervention, the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP), to increase activity in older adults by reducing emotional distress. The primary aim of the proposed study is to adapt a 5-session version of the UP for use with older adults reporting emotional distress and reduced engagement in daily activities and to develop a self-guided version of this intervention.

This aim will be accomplished in two phases. In Phase 1, patients will receive a short 5-session version of the UP via telehealth. At the end of treatment, they will provide feedback on the treatment, including any suggested changes, as well as suggestions for changing the treatment that might allow an individual to successfully complete it on their own. This information will be used to iteratively change the treatment and develop a self-guided version of the treatment.

In Phase 2, the study team will compare the therapist-delivered and self-guided versions of treatment to see if patients find them acceptable. In this phase, patients will be randomized to receive one of these two treatments.

DETAILED DESCRIPTION:
The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) is an optimal intervention to adapt for older adults to increase their engagement in daily activities. The UP is a type of cognitive behavioral therapy (CBT) with evidence base to reduce psychopathology, especially in transdiagnostic anxiety. As a transdiagnostic treatment, it can be applied across diagnostic categories to address a wide range of presenting problems. The UP is efficacious for anxiety, depression, and related emotional problems and has been used with older adults. The UP contains five core skills that are relevant to increasing activity engagement: Session 1 (Motivation & Psychoeducation about Emotions); Session 2 (Breaking down Emotions & Mindfulness); Session 3 (Cognitive Flexibility); Session 4 (Countering Emotion-Driven Behaviors); Session 5 (Exposure and Relapse Prevention).

Transdiagnostic treatments, like the UP, are advantageous for dissemination and implementation because they are adaptable and reduce clinician training burden. The UP has demonstrated adaptability for underserved patient populations and has been successfully abbreviated to meet the needs of unique patient populations. Further, it has been successfully delivered by clinicians without previous CBT experience, increasing its potential for dissemination. A five-session version of this treatment (UP-5) was developed that includes the core skills and showed acceptability in adults with acute suicide risk. The primary aim of this study is to adapt the UP-5 for use with older adults reporting emotional distress to increase their daily activity. Because research indicates the proportion of older adults who access and receive evidence-based treatments is low, the study team is proposing to develop therapist-delivered and self-guided versions of the treatment. Self-guided interventions may be ideal for older adults because they do not compete with other healthcare demands and they have the potential for significant public health impact for older adults where access to services is low. The secondary aim of this study is to compare the self-guided and therapist-delivered versions to begin identifying the minimum level of intervention needed to increase activity in older adults. This project is significant because it will produce an implementable, evidence-based treatment to increase access to evidence-based interventions designed to increase daily activity in older adults.

Phase 1. The purpose of Phase 1 was to adapt self-guided and therapist-delivered versions of the UP from the existing UP-5 using stakeholder feedback. The study used a successive cohort design and delivered the UP-5 to two cohorts of two patients (total of 4). One week after the fifth session, patients provided feedback about the treatment in exit interviews, which was used to develop and refine a self-guided version of the UP-5.

Phase 2. Phase 2 was a pilot randomized controlled trial comparing the adapted self-guided and therapist-delivered versions of the UP-5. Patients were randomized to complete one of these two treatments, 8 patients in each treatment arm. Therapist-delivered treatment was provided by telehealth via the study interventionist. All sessions were audio or video recorded so that a percentage could be rated for therapist adherence. Participants were provided with a pedometer to keep track of their step count throughout treatment. During each therapist-delivered treatment session, starting at session 2, the interventionist completed a Clinical Global Impressions-Improvement (CGI-I) rating and documented how much of the homework they thought the participant completed since the last session (0-100%). Outcomes were evaluated pre/post treatment and include measures of daily activity (PSFS), depression (PROMIS-depression), anxiety (PROMIS-anxiety), cognitive flexibility, experiential avoidance (BEAQ), and mindfulness (SMQ). Treatment satisfaction (Client-Satisfaction Questionnaire) and credibility and expectancy of improvement (CEIS) were evaluated post-treatment. The post-treatment visit was 1 week after completing self-guided or therapist-driven treatment. Five weeks after completing the final treatment session, measures and reporting of daily step count were collected remotely, one final time.

ELIGIBILITY:
Inclusion Criteria:

1. are age 65+
2. report moderate or higher emotional distress
3. report reduced engagement in daily activities
4. are willing to engage in telehealth.

Exclusion Criteria:

1. present with conditions requiring immediate prioritization (e.g., suicide attempt within past 6months, suicidal ideation with intent/plan, diagnosed with mania/bipolar I, psychosis)
2. are currently receiving psychotherapy
3. have been diagnosed with dementia or has significant concerns with memory as per online/phone screener
4. have changed their psychiatric medications in the past six weeks
5. cannot read
6. are blind
7. cannot speak English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrada Neacsiu, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be available on request and in compliance with IRB regulations.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.63 (5.975) | 69.5 (2.268) | 70.06 (4.404)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Patient Specific Functional Scale (PSFS) [Mean (Standard Deviation); unit: units on a scale] — The PSFS is a measure that can be used to quantify activity limitation and adapted to particular individuals and their functional status. Participants can include up to five activities, of which they rate their limitations on a 0-10 scale, where 0 corresponds to unable to perform and 10 corresponds to able to perform at the activity as well as usual . This scale is not necessarily designed for between subjects comparison of specific activities, but has been shown to be valid and responsive to change in musculoskeletal conditions within subjects.
  units on a scale | 4.1667 (1.03892) | 3.4583 (1.0974) | 3.8124 (1.095)
PROMIS Depression Total Score [Mean (Standard Deviation); unit: units on a scale] — The PROMIS Depression scale is measured on a scale from 8 to 40 with higher scores indicating more depression severity
  units on a scale | 24.3750 (7.2961) | 24.2500 (5.230) | 24.3125 (6.1179)
PROMIS Anxiety Total Score [Mean (Standard Deviation); unit: units on a scale] — PROMIS Anxiety measures anxiety severity on a scale from 7 to 35. Higher scores indicate more anxiety severity
  units on a scale | 23.7500 (2.8661) | 23.7500 (5.0071) | 23.7500 (3.9412)
Brief Experiential Avoidance Questionnaire (BEAQ) [Mean (Standard Deviation); unit: units on a scale] — The Brief Experiential Avoidance Questionnaire (BEAQ) is a 15-item self-report measure that assesses an individual's tendency to avoid or escape from unwanted internal experiences, such as uncomfortable emotions, thoughts, memories, or sensations. Higher scores represent more avoidance (range 15- 90)
  units on a scale | 48.50 (8.912) | 52.25 (11.411) | 50.38 (10.079)
Cognitive Flexibility Scale (CFS) [Mean (Standard Deviation); unit: score on a scale] — The cognitive flexibility scale ranges from 1 to 72, with higher scores indicating more flexibility in thinking than lower scores. It measures one's ability to adapt to changes in the environment.
  score on a scale | 56.6250 (7.1101) | 53.5000 (8.3666) | 55.0625 (7.6722)
Credibility and Expectancy Questionnaire (CEQ) [Mean (Standard Deviation); unit: score on a scale] — The CEQ is a six-item scale intended to measure patients' perceptions of a treatment's logicality and potential success with good evidence for validity and reliability. Participants rated each item on a scale from 1 to 9 ("not at all" - "very"). Items included how logical they perceived the treatment to be, how confident they were in the treatment, and how successful they thought the treatment was at improving emotional well-being and activity. A summary score is computed by averaging the answers, with higher scores indicating more credibility of the intervention (range 1-9).
  score on a scale | 5.7196 (1.1516) | 6.4218 (0.9424) | 6.1146 (1.0647)
PROMIS Physical Function Score [Mean (Standard Deviation); unit: score on a scale] — The PROMIS Physical Function Scale is an 8-item self-report examining difficulty with engaging in daily activities. Items are rated on a scale of 1-5 (unable to do -- can do without any difficulty), with lower scores representing more impairment in functioning. The scale ranges from 8 to 40.
  score on a scale | 32.7143 (6.5502) | 32.8889 (6.0919) | 32.8125 (6.0797)
Gait Speed (Mean of two trials) [Mean (Standard Deviation); unit: seconds] — The Short Physical Performance Battery (SPPB) is a performance-based assessment designed to evaluate lower extremity function in older adults(Guralnik et al., 1994). Performance was measured by a study team member through a virtual session before the first treatment session. Participants demarcate a length of three meters. Participants were instructed to walk this distance at their ordinary pace while the time was recorded to calculate their gait speed. Mean gait speed across two trials was calculated at each assessment.
  seconds | 4.0494 (1.4319) | 3.5794 (0.9460) | 3.8144 (1.1972)
Weekly Steps [Mean (Standard Deviation); unit: steps/week] — how many steps were taken per week recorded by a pedometer.
  steps/week | 3728.1786 (1572.4733) | 4098.9286 (2689.6560) | 3913.5536 (2136.9491)

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The CSQ is measured on a scale of 8-32, with higher scores indicating higher levels of treatment satisfaction
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post treatment | 30.5 (0.756) | 23.38 (4.779)
  1 Month Post treatment | 30.88 (1.642) | 25.25 (3.615)
Statistical Analysis 1: Comparison: Therapist Delivered Unified Protocol vs Self-Guided Unified Protocol; Test type: Superiority; p = .03, t-test, 2 sided; γ01 = .25 — analysis completed using the 1 week follow up data

2. Primary Outcome: Change in Patient Specific Functional Scale (PSFS)
Description: The PSFS is a measure that can be used to quantify activity limitation and adapted to particular individuals and their functional status. Participants can include up to five activities, of which they rate their limitations on a 0-10 scale, where 0 corresponds to unable to perform and 10 corresponds to able to perform at the activity as well as usual. This scale is not specifically designed for between-subjects comparisons of specific activities, but has been validated and shown to be sensitive to changes in musculoskeletal conditions within subjects. The scores represent changes from baseline at the reported follow-up periods
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Therapist Delivered Unified Protocol: This is a five session psychotherapy designed to help people with problems such as anxiety and depression. (duration: 5 weeks)
  Unified Protocol: Five session psychotherapy
- Self-Guided Unified Protocol: This is a five session treatment that patients can complete independently. (duration: 5 weeks)
  Unified Protocol: Five session psychotherapy
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post Treatment | 3.4167 (2.1658) | 3.2500 (1.6011)
  1 Month Post Treatment | 4.5833 (1.8148) | 4.2500 (1.7067)
Statistical Analysis 1: Comparison: Therapist Delivered Unified Protocol vs Self-Guided Unified Protocol; PSFS scores were analyzed using mixed-effects linear growth models with time, treatment condition, and their interaction as predictors. Random effects modeled variation in intercepts, slopes over time, and their covariance. Time was specified as a continuous variable, centered on the final observation date. The SG group served as the reference level for the treatment factor. Models were estimated in a Bayesian framework using default priors in the brms package; Test type: Other — The conditions were expected to be similar, and the primary interest of the analysis was changes over time across both groups; Bayesian framework — To estimate the mean improvement in PSFS across the entire sample, we calculated a posterior predictive distribution of within-person change scores between time fixed equal to 0 and equal to -1; Mean Difference (Final Values) = 3.40, 95% CI 2-sided [2.32 to 4.49]

3. Primary Outcome: Retention of Participants
Description: Retention of participants through completion of the study
Time Frame: 1 Month Post Treatment
Measure: Count of Participants; unit: Participants
Groups:
- Self-Guided Unified Protocol: This is a five session treatment that patients can complete independently.
  Unified Protocol: Five session psychotherapy (duration: 5 weeks)
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
Participants | 8 | 8

4. Secondary Outcome: Change in PROMIS-depression
Description: The PROMIS-depression is measured on a scale of 8-40, with higher scores indicating higher levels of depression. The scores represent changes from baseline at the reported follow up periods.
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post Treatment | -4.8750 (5.8417) | -1.875 (6.4901)
  1 Month Post Treatment | -6.2500 (5.1478) | -4.625 (4.5336)

5. Secondary Outcome: Change in PROMIS-anxiety
Description: The PROMIS-anxiety is measured on a scale of 7-35, with higher scores indicating higher levels of anxiety. The scores represent changes from baseline at the reported follow up periods.
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post Treatment | -4.000 (7.5024) | -1.1250 (4.7940)
  1 Month Post Treatment | -6.5000 (6.7612) | -5.375 (3.0677)

6. Secondary Outcome: Brief Experiential Avoidance Questionnaire (BEAQ).
Description: The Brief Experiential Avoidance Questionnaire (BEAQ) is a 15-item self-report measure that assesses an individual's tendency to avoid or escape from unwanted internal experiences, such as uncomfortable emotions, thoughts, memories, or sensations. Higher scores represent more avoidance (range 15- 90). The scores reported here represent changes from baseline at the reported follow up periods.
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
units on a scale
  1 Week Post | -11.8750 (12.4147) | -9.0000 (9.0396)
  1 Month Post | -11.2500 (16.2195) | -8.5000 (7.010)

7. Secondary Outcome: Cognitive Flexibility Scale (CFS)
Description: The Cognitive Flexibility Scale (CFS) measures one's ability to adapt in response to changes in environments and situations, on a range from 1 to 72. Higher scores on the CFS indicate greater cognitive flexibility. The scores represent changes from baseline at the reported follow-up periods. Therefore, a positive score represents an increase in cognitive flexibility from baseline.
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post Treatment | 4.37 (7.0495) | -2.0000 (10.7836)
  1 Month Post Treatment | 4.7500 (5.4182) | 6.8750 (8.4589)

8. Secondary Outcome: Southampton Mindfulness Questionnaire (SMQ)
Description: The SMQ ranges from 0 to 96, with higher scores indicating more mindfulness. The scores represent changes from baseline at the reported follow-up periods.
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post Treatment | 12.2857 (17.5187) | 7.1111 (16.1976)
  1 Month Post Treatment | 22.4286 (10.0155) | 14.3125 (17.1298)

9. Secondary Outcome: PROMIS Physical Function Score
Description: The PROMIS Physical Function Scale is an 8-item self-report examining difficulty with engaging in daily activities. Items are rated on a scale of 1-5 (unable to do -- can do without any difficulty), with lower scores representing more impairment in functioning. The scale ranges from 8 to 40. Here we present changes from baseline.
Time Frame: 1 week (post treatment), 1 month (post treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
score on a scale
  1 Week Post Treatment | 2.4286 (4.4293) | 2.3333 (2.5495)
  1 Month Post Treatment | 2.4286 (4.2370) | -0.7777 (4.9441)

10. Secondary Outcome: Gait Speed
Description: The Short Physical Performance Battery (SPPB) is a performance-based assessment designed to evaluate lower extremity function in older adults(Guralnik et al., 1994). The SPPB includes three components, but in this study, we utilized only the gait speed subtest. Performance was measured by a study team member through a virtual session at some point before the first treatment session and once again at the 1-week follow-up visit. Participants were mailed necessary materials, including measuring tape and black tape, to demarcate a length of three meters. Participants were instructed to walk this distance at their ordinary pace while the time was recorded to calculate their gait speed. Mean gait speed across two trials was calculated at each assessment.
Time Frame: Baseline (1 week before treatment), 1 week post treatment
Population: There were two participants for whom data was not collected due to administrative error at 1 week post treatment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
seconds
  1 week before treatment (baseline) | 4.049 (1.4319) | 3.579 (0.9460)
  1 Week Post Treatment: number analyzed (Participants) | 6 | 8
  1 Week Post Treatment | 3.8983 (1.1390) | 3.6650 (0.9939)

11. Secondary Outcome: Weekly Steps
Description: average for each condition of total weekly steps taken by study participants measured on a pedometer
Time Frame: at baseline (i.e., the week before session 1 of treatment), during each of the four remaining therapy weeks (session 1--> session 2; 2--> 3; 3-->4; 4--> 5), the week following treatment, the week following a month after treatment ended.
Population: data missing (not submitted) for 2 participants at the 1 month follow up and 1 participant at the 1 week follow up.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
steps
  Baseline | 26097.25 (11007.31312) | 28692.5 (18827.59205)
  Week 1 in treatment | 24075.25 (13210.29827) | 30716.8750 (21695.55241)
  Week 2 in treatment | 26809.3750 (14895.31271) | 32359.7500 (20783.19429)
  Week 3 in treatment | 30367.875 (24098.26813) | 43975.50 (36506.15559)
  Week 4 in treatment | 30933.3750 (20550.41131) | 35602.000 (24011.11186)
  The week after treatment: number analyzed (Participants) | 7 | 8
  The week after treatment | 26254.7143 (17190.26649) | 40353.6250 (26573.42281)
  the week following a month after treatment: number analyzed (Participants) | 8 | 6
  the week following a month after treatment | 29993.25 (23367.89734) | 38454.8333 (35403.89371)

12. Secondary Outcome: Credibility and Expectancy Score
Description: The CEQ (Devilly & Borkovec, 2000) is a six-item scale intended to measure patients' perceptions of a treatment's logicality and potential success with good evidence for validity and reliability. At intake, we administered a 6-item adaptation, assessing how logical the UP protocol sounded before being administered and expectations about how effective the treatment would be in reducing distress. We then administered a 5-item adapted version of this questionnaire at one-week and one-month follow-up visits. Participants rated each item on a scale from 1 to 9 ("not at all" - "very"). Items included how logical they perceived the treatment to be, how confident they were in successfully using the strategies presented and recommending it to a friend, and how successful they thought the treatment was at improving emotional well-being and activity levels. A summary score is computed by averaging the answers, with higher scores indicating more credibility of the intervention (range 1-9).
Time Frame: one week after treatment, one month after treatment
Population: Mean scores
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
Number analyzed (Participants) | 8 | 8
units on a scale
  One week after treatment | 8.3000 (0.8751) | 6.550 (1.4570)
  One month after treatment | 7.8250 (1.0222) | 6.775 (1.317)

13. Secondary Outcome: Percent of Adherent Sessions Completed in the Therapist Delivered Arm of the Study.
Description: A rater trained by the PI scored 35% of therapist-driven sessions. Each session was rated using yes/no answers for 12 different domains . An overall computed score captured how many domains were coded as yes in the particular session. The session duration needed to be at least 30 minutes for the session to be considered adherent. In addition, each session was rated for adequacy using 5 items that assessed the therapist's level of engagement and ability to manage the session on a 0-5 scale("Poor" to "Excellent"). These items were averaged. We computed a binary yes/no score that captured whether the session adhered to the protocol. To be adherent, a session needed to include at least 10/12 elements and have an average adequacy rating of at least 3/5. Adherence was not measured in the self-help group because the therapist did not deliver any direct intervention in this group. We present the percentage of sessions coded as adherent from a random selection of videotaped sessions.
Time Frame: End of the 5 week-treatment for all participants, approximately 2 months
Measure: Number; unit: percent of sessions coded at adherence
Units Other Than Participants: Number of sessions
Arm/Group | Therapist Delivered Unified Protocol
Number analyzed (Participants) | 8
Number analyzed (Number of sessions) | 14
percent of sessions coded at adherence | 92.3

ADVERSE EVENTS:
Time Frame: Reports of adverse events were self reported by participants during their enrollment in the study. (weeks 0 - 12 from intake)
Arm/Group | Therapist Delivered Unified Protocol | Self-Guided Unified Protocol
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 5/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapist Delivered Unified Protocol (N=8) | Self-Guided Unified Protocol (N=8)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated to study procedures. Intermittent.
Broken Wrist/Ribs/Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Secondary to accidental fall. Unrelated to study. Ongoing.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapist Delivered Unified Protocol (N=8) | Self-Guided Unified Protocol (N=8)
Respiratory Virus (General disorders) | 1 (1) | 0 (0) — Unrelated to study procedures.Resolved without sequelae.
Twisted Ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Secondary to fall. Unrelated to study. Persistent.
Accidental Fall (General disorders) | 1 (1) | 0 (0) — Single event. Unrelated to study. Resolved without sequelae.
Fatigue post oral surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Unrelated to study. Resolved without sequelae.
Pulled Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Strain in muscle in back. Unrelated to study. Resolved without sequelae
Broken Wrist (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to study. Persistent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04837521/Prot_001.pdf
  • Statistical Analysis Plan (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT04837521/SAP_002.pdf
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04837521/ICF_000.pdf